CLINICAL TRIAL: NCT00468299
Title: Treatment of Early Pregnancy Failure
Brief Title: MiMi: A Randomized Trial of Mifepristone and Misoprostol for Treatment of Early Pregnancy Failure
Acronym: MiMi
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: Boston University (Other)
Responsible Party: Sarah Betstadt, MD, University of Rochester Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-25999
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-06

CONDITIONS: Early Pregnancy Failure; Miscarriage; Fetal Demise; Anembryonic Pregnancy
Keywords: early; pregnancy; failure; mifepristone; misoprostol; buccal; miscarriage; fetal; demise; anembryonic; progesterone
MeSH Terms: conditions — Abortion, Spontaneous; Fetal Death | interventions — Misoprostol; Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol and placebo (Active Comparator): Women in this arm receive placebo and misoprostol 800 mcg buccally
  Interventions: Drug: Misoprostol and placebo
- Mifepristone and misoprostol (Experimental): Womwn in this group receive mifepristone 200 mg orally and misoprostol 800 mcg buccally
  Interventions: Drug: Mifepristone and misoprostol

INTERVENTIONS:
Drug: Misoprostol and placebo — Women in this group receive 800 mcg misoprostol plus a placebo
  Arms: Misoprostol and placebo
Drug: Mifepristone and misoprostol — This group receives mifepristone 200 mg orally; followed by 800 mcg misoprostol bucally
  Arms: Mifepristone and misoprostol

SUMMARY:
The purpose of this study is to compare two combinations of drugs (mifepristone and misoprostol versus placebo and misoprostol) used for medical treatment for early pregnancy failure. We will compare the two combinations of medications to see which combination makes miscarriage happen faster. We hypothesize that there will be no difference in time to complete miscarriage between the two groups.

DETAILED DESCRIPTION:
The optimal method of treating Early Pregnancy Failure (EPF) is not certain. For many years, surgical management of EPF was the only treatment option. Now there are multiple studies demonstrating the effectiveness of misoprostol for treating EPF. Most of the studies investigating medical treatment of EPF have evaluated efficacy at one week. We have found that many women do not want to wait for one week for an outcome of their medical treatment, and want resolution sooner. This has hampered the widespread utilization of medical therapy in our institution.

We propose a regimen of medical treatment for EPF with expeditious follow-up. We want to demonstrate the relative efficacy of two medication regimens for treatment of EPF by performing a randomized trial. One regimen will be 800μg buccal misoprostol alone and the other regimen will be 200mg mifepristone, orally, in addition to 800μg buccal misoprostol, simultaneously. The primary outcome will be complete abortion rates 24hours after medication administration. We hypothesize that mifepristone will not improve complete abortion rates at 24hrs.

Secondary outcomes include rates of abortion by medical treatment at one week, the indications for surgical intervention, relationship of progesterone levels and type of pregnancy failure to outcomes in the two groups. Another secondary objective is to assess satisfaction with the treatment process at the conclusion of pregnancy termination, and 3 weeks after the beginning of the process.

The majority of studies investigating medical treatment of EPF use vaginal misoprostol, but buccal use is increasing. We will use buccal misoprostol, which is widely used at our institution. We will assess the efficacy of this route of administration as well as assess patient acceptability of this method.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yrs, able to read and write English
* Intrauterine gestations with anembryonic sac between 10 and 45mm or
* 10-15mm sac with no growth in three days or other radiologic signs of abnormal pregnancy such as irregular sac or debris within the gestational sac
* An embryonic pole <30mm with no cardiac activity

Exclusion Criteria:

* Intrauterine gestations with CRL <5mm or >30mm without cardiac activity
* Incomplete abortion as defined as open cervix and large amount of cramping/bleeding
* Hemodynamic instability and/or heavy vaginal bleeding
* Hemoglobin less than or equal to 8
* Inability to follow-up (ie, lack of transportation or access to telephone)
* Bleeding disorder or taking anticoagulants
* Prior medical or surgical treatment of the current pregnancy
* Obvious Infection
* Active Lactation
* Allergy to mifepristone or misoprostol
* Chronic corticosteroid use
* Severe gastrointestinal disease (e.g inflammatory bowel disease, severe gastritis)

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Betstadt, MD, Principal Investigator — Boston University; Olivera Vragovic, MBA, Study Director — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bagratee JS, Khullar V, Regan L, Moodley J, Kagoro H. A randomized controlled trial comparing medical and expectant management of first trimester miscarriage. Hum Reprod. 2004 Feb;19(2):266-71. doi: 10.1093/humrep/deh049. PMID 14747165
- [Background] Creinin MD, Schwartz JL, Guido RS, Pymar HC. Early pregnancy failure--current management concepts. Obstet Gynecol Surv. 2001 Feb;56(2):105-13. doi: 10.1097/00006254-200102000-00024. PMID 11219590
- [Background] Lelaidier C, Saint-Mleux CB, Fernandez H, Bourget P, Frydman R. [Embryo expulsion induction in first trimester miscarriages. Use of mifepristone (RU 486) in a double blind prospective randomized study]. Contracept Fertil Sex. 1993 Jun;21(6):505-8. French. PMID 7920940
- [Background] Lister MS, Shaffer LE, Bell JG, Lutter KQ, Moorma KH. Randomized, double-blind, placebo-controlled trial of vaginal misoprostol for management of early pregnancy failures. Am J Obstet Gynecol. 2005 Oct;193(4):1338-43. doi: 10.1016/j.ajog.2005.05.010. PMID 16202723
- [Background] Meckstroth KR, Whitaker AK, Bertisch S, Goldberg AB, Darney PD. Misoprostol administered by epithelial routes: Drug absorption and uterine response. Obstet Gynecol. 2006 Sep;108(3 Pt 1):582-90. doi: 10.1097/01.AOG.0000230398.32794.9d. PMID 16946218
- [Background] Middleton T, Schaff E, Fielding SL, Scahill M, Shannon C, Westheimer E, Wilkinson T, Winikoff B. Randomized trial of mifepristone and buccal or vaginal misoprostol for abortion through 56 days of last menstrual period. Contraception. 2005 Nov;72(5):328-32. doi: 10.1016/j.contraception.2005.05.017. Epub 2005 Aug 9. PMID 16246656
- [Background] Nielsen S, Hahlin M, Platz-Christensen JJ. Unsuccessful treatment of missed abortion with a combination of an antiprogesterone and a prostaglandin E1 analogue. Br J Obstet Gynaecol. 1997 Sep;104(9):1094-6. doi: 10.1111/j.1471-0528.1997.tb12075.x. PMID 9307543
- [Background] Schaff EA, DiCenzo R, Fielding SL. Comparison of misoprostol plasma concentrations following buccal and sublingual administration. Contraception. 2005 Jan;71(1):22-5. doi: 10.1016/j.contraception.2004.06.014. PMID 15639067
- [Background] Stockheim D, Machtinger R, Wiser A, Dulitzky M, Soriano D, Goldenberg M, Schiff E, Seidman DS. A randomized prospective study of misoprostol or mifepristone followed by misoprostol when needed for the treatment of women with early pregnancy failure. Fertil Steril. 2006 Oct;86(4):956-60. doi: 10.1016/j.fertnstert.2006.03.032. PMID 17027362
- [Background] Tang OS, Schweer H, Seyberth HW, Lee SW, Ho PC. Pharmacokinetics of different routes of administration of misoprostol. Hum Reprod. 2002 Feb;17(2):332-6. doi: 10.1093/humrep/17.2.332. PMID 11821273
- [Background] Trinder J, Brocklehurst P, Porter R, Read M, Vyas S, Smith L. Management of miscarriage: expectant, medical, or surgical? Results of randomised controlled trial (miscarriage treatment (MIST) trial). BMJ. 2006 May 27;332(7552):1235-40. doi: 10.1136/bmj.38828.593125.55. Epub 2006 May 17. PMID 16707509
- [Background] Wagaarachchi PT, Ashok PW, Smith NC, Templeton A. Medical management of early fetal demise using sublingual misoprostol. BJOG. 2002 Apr;109(4):462-5. doi: 10.1111/j.1471-0528.2002.01075.x. PMID 12013170
- [Background] Wagaarachchi PT, Ashok PW, Narvekar N, Smith NC, Templeton A. Medical management of early fetal demise using a combination of mifepristone and misoprostol. Hum Reprod. 2001 Sep;16(9):1849-53. doi: 10.1093/humrep/16.9.1849. PMID 11527887
- [Background] Zhang J, Gilles JM, Barnhart K, Creinin MD, Westhoff C, Frederick MM; National Institute of Child Health Human Development (NICHD) Management of Early Pregnancy Failure Trial. A comparison of medical management with misoprostol and surgical management for early pregnancy failure. N Engl J Med. 2005 Aug 25;353(8):761-9. doi: 10.1056/NEJMoa044064. PMID 16120856
- [Background] Zieman M, Fong SK, Benowitz NL, Banskter D, Darney PD. Absorption kinetics of misoprostol with oral or vaginal administration. Obstet Gynecol. 1997 Jul;90(1):88-92. doi: 10.1016/S0029-7844(97)00111-7. PMID 9207820

RESULTS

PARTICIPANT FLOW:
Groups:
- Misoprostol and Placebo: Women in this groups received misoprostol (800 mcg buccally) plus a placebo for treatment of early pregnancy failure.
- Mifepristone and Misoprostol: Women in this group received mifepristone 200 mg orally followed by misoprostol 800 mcg buccally
Period: Overall Study
Arm/Group | Misoprostol and Placebo | Mifepristone and Misoprostol
Started | 9 | 8
Completed | 9 | 7
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol and Placebo | Mifepristone and Misoprostol | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28 (4) | 29 (4) | 28 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Women With Complete Abortion 24-48hrs After Receiving Medical Treatment for Early Pregnancy Failure.
Time Frame: 24-48 hrs
Measure: Number; unit: participants
Arm/Group | Misoprostol and Placebo | Mifepristone and Misoprostol
Number analyzed (Participants) | 9 | 8
participants | 5 | 5

2. Secondary Outcome: Complete Abortion at One Week
Description: Complete abortion at one week; uterus demonstrated to be empty on transvaginal ultrasound
Time Frame: 3 weeks
Population: Per protocol
Measure: Number; unit: participants
Groups:
- Misoprostol and Placebo: Women received a placebo followed by misoprostol 800 mcg buccally
- Mifepristone and Misoprostol: Women received mifeppristone 200 mg orally followed ny misoprostol 800 mcg buccally
Arm/Group | Misoprostol and Placebo | Mifepristone and Misoprostol
Number analyzed (Participants) | 9 | 8
participants | 6 | 7

ADVERSE EVENTS:
Arm/Group | Misoprostol and Placebo | Mifepristone and Misoprostol
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
The study was terminated because of poor enrollment. Few eligible women were referred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No